CLINICAL TRIAL: NCT04269395
Title: A Double-blind, Multicenter, Long-term Follow-up Study to Assess Recurrence of Actinic Keratosis in Subjects Treated With Methyl Aminolevulinate Hydrochloride (MAL) 16.8% Cream (CD06809-41) or Vehicle Cream in the Treatment of Thin and Moderately Thick, Non-hyperkeratotic, Non-pigmented Actinic Keratosis of the Face and Scalp When Using Daylight Photodynamic Therapy (DL-PDT), for Subjects Achieving Complete Response of Treated Lesions at Final Visit in Study RD.06.SPR.112199
Brief Title: A Study to Assess Recurrence of Actinic Keratosis in Participants Treated With Methyl Aminolevulinate Hydrochloride Cream or Vehicle Cream Who Achieved Complete Response to Treated Lesions in Earlier Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early as per Sponsor's decision
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RD.06.SPR.115230
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Keratosis, Actinic
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAL Cream Arm (Active Comparator): Participants who completed the study RD.06.SPR.112199 (NCT04085367) and achieved complete response of all treated lesions at the final visit of the active cream group, will continue for long-term follow-up to evaluate recurrence of AKs in this study.
  Interventions: Drug: MAL Cream
- Vehicle Cream Arm (Placebo Comparator): Participants who completed the study RD.06.SPR.112199 (NCT04085367) and achieved complete response of all treated lesions at the final visit in the vehicle cream group, will continue for long-term follow-up to evaluate recurrence of AKs in this study.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: MAL Cream — No intervention will be administered as a part of this study. Participants who received MAL cream in RD.06.SPR.112199 study will be rolled over in the study.
  Other Names: CD06809-41
  Arms: MAL Cream Arm
Drug: Vehicle cream — No intervention will be administered as a part of this study. Participants who received vehicle cream in RD.06.SPR.112199 study and achieved complete response, will be rolled over in the study.
  Arms: Vehicle Cream Arm

SUMMARY:
The primary purpose for this study is to assess recurrence of Actinic Keratosis in participants achieving complete response treated in earlier study.

DETAILED DESCRIPTION:
This is a double-blind, multicenter, long-term follow-up study. The primary purpose of this study is to assess recurrence of Actinic Keratosis in participants treated with Methyl aminolevulinate hydrochloride (MAL) 16.8 percent (%) cream (CD06809-41) or vehicle cream in the treatment of thin and moderately thick, non-hyperkeratotic, non-pigmented actinic keratosis of the face and scalp when using daylight photodynamic therapy (DL-PDT), for participants achieving complete response of treated lesions at Final Visit in Study RD.06.SPR.112199 (NCT04085367).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed earlier study RD.06.SPR.112199 (NCT04085367) and achieved complete response at last visit
* Participants fully understand and sign an informed consent form (ICF) before any study procedure begins
* Participants willing and able to perform all study protocol requirements

Exclusion Criteria:

* Participants developing or experiencing any condition that may not be safe for them or not compliant will be excluded
* Pertinent not compliant with study conditions or PI instructions during the earlier study - Lumexia Ph 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (49):
  - Galderma Investigational Site (Site#8447), Fort Smith, Arkansas
  - Galderma Investigational Site (Site#8577), Encinitas, California
  - Galderma Investigational Site (Site#8636), Fountain Valley, California
  - Galderma Investigational Site (Site#8224), Fremont, California
  - Galderma Investigational Site (Site#8778), Denver, Colorado
  - Galderma Investigational Site (Site#8440), Greenwood Village, Colorado
  - Galderma Investigational Site (Site#8479), Bradenton, Florida
  - Galderma Investigational Site (Site#8769), Lake Worth, Florida
  - Galderma Investigational Site (8770), Lehigh Acres, Florida
  - Galderma Investigational Site (Site#8765), North Miami Beach, Florida
  - Galderma Investigational Site (Site#8734), Pembroke Pines, Florida
  - Galderma Investigational Site (Site#8529), Sanford, Florida
  - Galderma Investigational Site (Site#8126), West Palm Beach, Florida
  - Galderma Investigational Site (Site#8667), Columbus, Georgia
  - Galderma Investigational Site (Site#8755), Boise, Idaho
  - Galderma Investigational Site, Boise, Idaho
  - Galderma Investigational Site (Site#8838), Darien, Illinois
  - Galderma Investigational Site (Site#8724), Louisville, Kentucky
  - Galderma Investigational Site (Site#8208), Beverly, Massachusetts
  - Galderma Investigational Site (Site#8574), Clarkston, Michigan
  - Galderma Investigational Site (Site#8757), Saint Joseph, Michigan
  - Galderma Investigational Site, Edina, Minnesota
  - Galderma Investigational Site, St Louis, Missouri
  - Galderma Investigational Site (Site#8048), Omaha, Nebraska
  - Galderma Investigational Site 9Site#8420), Portsmouth, New Hampshire
  - Galderma Investigational Site (Site#8759), Albuquerque, New Mexico
  - Galderma Investigational Site, Brooklyn, New York
  - Galderma Investigational Site, New York, New York
  - Galderma Investigational Site (Site#8566), Charlotte, North Carolina
  - Galderma Investigational Site (Site#8595), Dublin, Ohio
  - Galderma Investigational Site (Site#8212), Portland, Oregon
  - Galderma Investigational Site, Philadelphia, Pennsylvania
  - Galderma Investigational Site, Pittsburgh, Pennsylvania
  - Galderma Investigational Site, Sugarloaf, Pennsylvania
  - Galderma Investigational Site (Site#8777), Charleston, South Carolina
  - Galderma Investigational Site (Site#8207), Nashville, Tennessee
  - Galderma Investigational Site (Site#8076), Austin, Texas
  - Galderma Investigational Site (Site#8139), College Station, Texas
  - Galderma Investigational Site (Site#8664), Frisco, Texas
  - Galderma Investigational Site (Site#8576), Houston, Texas
  - Galderma Investigational Site (Site#8546), Pflugerville, Texas
  - Galderma Investigational Site (Site#8761), Salt Lake City, Utah
  - Galderma Investigational Site (Site#8672), Salt Lake City, Utah
  - Galderma Investigational Site (Site#8776), St. George, Utah
  - Galderma Investigational Site (Site#8057), Lynchburg, Virginia
  - Galderma Investigational Site (Site#8779), Seattle, Washington
  - Galderma Investigational Site (Site#8760), Spokane, Washington
  - Galderma Investigational Site 2(Site#8039), Spokane, Washington
  - Galderma Investigational Site (Site#8725), Morgantown, West Virginia
- Galderma Investigational Site (Site#8231), Aibonito, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 study centers in United States from 7 April 2020 to 1 September 2021. Participants who completed study RD.06.SPR.112199 (NCT04085367) and achieved complete response (CR) of all treated Actinic Keratosis (AKs) lesions at final visit of treatment, were continued to be followed in this for long-term follow-up (LTFU) study to assess recurrence.
Pre-assignment Details: 125 participants (87 in Methyl aminolevulinate hydrochloride (MAL) 16.8% cream group and 38 in vehicle cream group) from main study RD.06.SPR.112199 were enrolled and treated in this study. Study was terminated early as in main study, primary analysis did not show superiority of MAL 16.8% cream with DL-PDT over vehicle cream with DL-PDT as of participant complete response (CR), and the sponsor decided not to apply for marketing authorization for the MAL 16.8% cream in combination with DL-PDT.
Groups:
- MAL Cream Arm: Participants who completed the study RD.06.SPR.112199 (NCT04085367) and achieved complete response of all treated lesions at the final visit of the active cream group (MAL), continued for long-term follow-up to evaluate recurrence of AKs in this study. No treatment was given to participants in this study.
- Vehicle Cream Arm: Participants who completed the study RD.06.SPR.112199 (NCT04085367) and achieved complete response of all treated lesions at the final visit in the vehicle cream group, continued for long-term follow-up to evaluate recurrence of AKs in this study. No treatment was given to participants in this study.
Period: Overall Study
Arm/Group | MAL Cream Arm | Vehicle Cream Arm
Started | 87 | 38
Completed | 73 | 28
Not Completed | 14 | 10
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study terminated by Sponsor | 13 | 10

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all enrolled participants and was to be used for all efficacy and safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | MAL Cream Arm | Vehicle Cream Arm | Total
Number analyzed (Participants) | 87 | 38 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (8.88) | 66.8 (8.89) | 68.5 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 58 | 13 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87 | 38 | 125
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Type I = White; very fair, red or blonde hair blue eyes; freckles; Always burns, never tans Type II = White, fair, red or blond hair; blue, hazel or green eyes; Usually burns, tans with difficulty Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily Type VI = Black; Never burns, tans very easily.
  Participants
    Type I | 6 | 1 | 7
    Type II | 43 | 16 | 59
    Type III | 35 | 19 | 54
    Type IV | 3 | 2 | 5
    Type V | 0 | 0 | 0
    Type VI | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Any (>=1) Cleared Treated AK Lesions at Week 54
Description: Participants with recurrence are defined as the participants with recurrence of any (greater than and equal to [>=] 1) cleared treated AK lesions. Number of participants with recurrence of any (>=1) cleared treated AK lesions at Week 54 was reported.
Time Frame: At Week 54
Population: Safety population consisted of all enrolled participants and was to be used for all efficacy and safety analyses. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | MAL Cream Arm | Vehicle Cream Arm
Number analyzed (Participants) | 75 | 30
Participants | 30 | 12

2. Secondary Outcome: Percent Recurrence of Cleared Treated AK Lesions at Week 28 and Week 54
Description: Recurrence is defined as the percentage of recurrence of cleared treated lesions. Percent recurrence of cleared treated actinic keratosis lesions at Week 28 and Week 54 was reported.
Time Frame: At Week 28 and Week 54
Population: Safety population consisted of all enrolled participants and was to be used for all efficacy and safety analyses. Screen failures were not to be included in the safety population. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percent recurrence
Arm/Group | MAL Cream Arm | Vehicle Cream Arm
Number analyzed (Participants) | 81 | 38
Percent recurrence
  At Week 28 | 6.91 (14.875) | 7.50 (16.154)
  At Week 54: number analyzed (Participants) | 75 | 30
  At Week 54 | 10.46 (15.692) | 12.72 (20.669)

3. Secondary Outcome: Number of Participants With Recurrence of Any (>=1) Cleared Treated AK Lesions at Week 28
Description: Participants with recurrence are defined as the participants with recurrence of any (greater than and equal to [>=] 1) cleared treated AK lesions. Number of participants with recurrence of any (>=1) cleared treated AK lesions at Week 28 was reported.
Time Frame: At Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MAL Cream Arm | Vehicle Cream Arm
Number analyzed (Participants) | 81 | 38
Participants | 19 | 8

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 54
Description: Safety population consisted of all enrolled participants and was to be used for all efficacy and safety analyses.
Arm/Group | MAL Cream Arm | Vehicle Cream Arm
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/38
Other Adverse Events (participants affected / at risk) | 22/87 | 11/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAL Cream Arm (N=87) | Vehicle Cream Arm (N=38)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 12 | 5
Androgenetic Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Application site erythema (General disorders) | 3 | 1
Application site atrophy (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 0
Corona virus infection (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This LTFU study was terminated early by the Sponsor because in the main study RD.06.SPR.112199, the primary analysis did not show superiority of MAL 16.8% cream with DL-PDT over vehicle cream with DL-PDT in terms of participant complete response (CR), and the sponsor decided not to apply for marketing authorization for the MAL 16.8% cream in combination with DL-PDT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT04269395/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT04269395/SAP_001.pdf